CLINICAL TRIAL: NCT03717389
Title: The Prevalence of Soft Tissue Calcifications in the Head and Neck Region Using CBCT Among Egyptian Population: Observational Cross Sectional Study
Brief Title: The Prevalence of Soft Tissue Calcifications in the Head and Neck Region Using CBCT Among Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maha Samy Elhadidy (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Maha Samy Elhadidy, postgraduate student, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 2371987
Record Dates: First submitted 2018-10-18; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Oral Soft Tissue Conditions
Keywords: prevalence; soft tissue calcification in head and neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: presence of soft tissue calcification in head and neck — soft tissue calcifications of the head and neck region in the Egyptian population

SUMMARY:
Prevalence of soft tissue calcifications in the head and neck region is not clearly studied in the Egyptian population.

Determining the incidence of these calcifications can improve the knowledge of dental practitioners and allow such practitioners to initiate proper diagnostic. And if patients need treatment they can start early by the right therapy to stop the.

The aim of this research is to detect and quantify the prevalence of the soft tissue calcifications by cone beam computed tomography (CBCT) images of the head and neck region in the Egyptian population.

DETAILED DESCRIPTION:
Calcification of various structures located in the head and neck region are reported in patients seeking dental care.

Although most of the soft tissue calcification within the head and neck region might not be accompanied by clinical symptoms; the investigators should not assume that their detection do not has a strong clinical significance .

Some soft tissue calcification may suggest the presence of a systemic condition and may cause threatening consequences .

Understanding of the nature of soft tissue calcification in the head and neck helps in proper diagnosis of these calcification and in turn taking the right decision of asking for further investigation; referral or do nothing .

Also; many of the structures in the head and neck region are in close proximity to one another which makes identification and localization difficult and this may lead to false diagnosis .

CBCT is a valuable imaging modality to overcome this difficulty. The data collection for this study will be obtained from the data base available at the Oral and Maxillofacial Radiology department at the faculty of dentistry -Cairo university

The following information will be recorded for each patient by :

1. Age of the patient at the time of the scan . 2. Sex (male or female). 3. Type of the scan (mandible only, maxilla and mandible, and full scan).

* Assessment will be made for the following;

  1. Presence or absence of calcification.
  2. Type of calcification present (or what is this soft tissue structure).
  3. Side (i.e. unilateral or bilateral and what side) .
  4. Single or multiple occurring.
* During assessing the CBCT images; neither clinical information nor demographic data of the patients will be available to any of the two radiologists.
* Then inter-observational and intra-observational variability between the observers will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans of 0.2 mm Voxel size will be included
* Scans that clearly show mandible only; maxilla only; maxilla and mandible or whole face will be included.
* Patients age 10-80 years old .

Exclusion Criteria:

* • Images with (Field Of View) show only one tooth or teeth.

  * Images of poor quality will be excluded.
  * Images showing artifacts caused by metallic implants or osteosynthesis plates.
  * Images subjected to patient movement during acquisition will be excluded also.

Ages: 10 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 350 CBCT scans belonging to Egyptian individuals who had CBCT examination as part of their dental treatment planning during the years 2017-2018-2019.from the data base available at the Oral and Maxillofacial Radiology department at the faculty of dentistry -Cairo university
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
what is percent of participants having soft tissue calcification among the whole population included"whether males or females" | the participants will be assessed 2 times at 2 weeks interval
  percentage%

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khojastepour L, Haghnegahdar A, Sayar H. Prevalence of Soft Tissue Calcifications in CBCT Images of Mandibular Region. J Dent (Shiraz). 2017 Jun;18(2):88-94. PMID 28620632
- [Background] Caglayan F, Sumbullu MA, Miloglu O, Akgul HM. Are all soft tissue calcifications detected by cone-beam computed tomography in the submandibular region sialoliths? J Oral Maxillofac Surg. 2014 Aug;72(8):1531.e1-6. doi: 10.1016/j.joms.2014.04.005. Epub 2014 Apr 13. PMID 25037186
- [Background] Guarda-Nardini L, Piccotti F, Ferronato G, Manfredini D. Myositis ossificans traumatica of the temporalis muscle: a case report and diagnostic considerations. Oral Maxillofac Surg. 2012 Jun;16(2):221-5. doi: 10.1007/s10006-011-0293-6. Epub 2011 Sep 22. PMID 21938392
- [Background] Lewis DA, Brooks SL. Cartoid artery calcification in a general dental population: a retrospective study of panoramic radiographs. Gen Dent. 1999 Jan-Feb;47(1):98-103. PMID 10321159